CLINICAL TRIAL: NCT06337734
Title: The Effect of an Artificial Intelligence-based, Autonomous, Digital Health Intervention Using Precise Lifestyle Guidance on Blood Pressure in Adults With Hypertension: Single-Arm Nonrandomized Trial
Brief Title: An Artificial Intelligence-Assisted Digital Health Lifestyle Intervention for Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sujit Dey, Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-Driven Lifestyle Coaching Group (Experimental)
  Interventions: Behavioral: AI-Driven Lifestyle Coaching Program

INTERVENTIONS:
Behavioral: AI-Driven Lifestyle Coaching Program — The intervention provides participants with automated and personalized lifestyle recommendations involving a sophisticated analytics engine using advanced statistics and machine learning.

SUMMARY:
This study evaluates the impact of a fully digital, autonomous, and artificial intelligence (AI)-driven lifestyle coaching program on managing blood pressure (BP) among adults diagnosed with hypertension. Participants received a BP monitor and a wearable activity tracker to facilitate data collection. This data, along with responses from a questionnaire mobile app, were analyzed by an automated analytics engine employing statistical and machine learning techniques. The program delivered tailored lifestyle coaching directly to participants through a mobile app, aiming for precise and effective BP management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Stage 2 hypertension based on their most recent clinical measurement (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg per the 2017 American College of Cardiology/American Heart Association guidelines)
* Speaking and reading English
* Having an Apple iPhone 6s or later, or an Android phone running Android 8.0 or later

Exclusion Criteria:

* Self-reported diagnosis of coronary heart disease, medical condition or other physical problem necessitating special attention in an exercise program (e.g., cancer, eating disorder, uncontrolled diabetes)
* Current participation in a lifestyle modification program or research study
* Self-report of being currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Average change in systolic blood pressure (SBP) from baseline to 12 weeks | 12 weeks
Average change in diastolic blood pressure (DBP) from baseline to 12 weeks | 12 weeks
Average change in SBP from baseline to 24 weeks | 24 weeks
Average change in DBP from baseline to 24 weeks | 24 weeks
Percent change of participants with controlled BP (SBP<130 and DBP<80) from baseline to 12 weeks | 12 weeks
Percent change of participants with controlled BP (SBP<130 and DBP<80) from baseline to 24 weeks | 24 weeks
Percent change of participants with Stage 2 Hypertension (SBP≥140 or DBP≥90) from baseline to 12 weeks | 12 weeks
Percent change of participants with Stage 2 Hypertension (SBP≥140 or DBP≥90) from baseline to 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Average weekly percentage of active participants measuring their BP | 24 weeks
Average weekly percentage of active participants syncing their wearable | 24 weeks
Average weekly percentage of active participants answering the mobile app questionnaire | 24 weeks
Number of manual clinician outreaches based on the escalation rules set for the study | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Leitner J, Chiang PH, Agnihotri P, Dey S. The Effect of an AI-Based, Autonomous, Digital Health Intervention Using Precise Lifestyle Guidance on Blood Pressure in Adults With Hypertension: Single-Arm Nonrandomized Trial. JMIR Cardio. 2024 May 28;8:e51916. doi: 10.2196/51916. PMID 38805253